CLINICAL TRIAL: NCT04205136
Title: Spironolactone to Improve Apnea and Cardiovascular Markers in Obstructive Sleep Apnea Patients With Cardiovascular Disease Who Are Non-Adherent With Positive Airway Pressure: A Randomized Placebo-Controlled Pilot Trial
Brief Title: Spironolactone to Improve Apnea and Cardiovascular Markers in Obstructive Sleep Apnea Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Was on hold due to Covid then we were not able to initiate the funding again after such a long hold and loss of team members.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Louise O'Brien, Research Associate Professor, Neurology, Research Associate Professor, Obstetrics and Gynecology, Medical School and Associate Research Scientist, Dentistry, Department of Oral and Maxillofacial Surgery, School of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUM00147375
Record Dates: First submitted 2019-12-11; First posted 2019-12-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Spironolactone; Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: The researchers will do a trial of spironolactone in 30 obstructive sleep apnea (OSA) patients with cardiovascular disease who are non-adherent with Positive Airway Pressure (PAP) therapy.
Who Masked: Participant, Investigator
Masking Description: Both groups will receive treatment as usual for obstructive sleep apnea. Spironolactone and placebo will be prescribed by one of the study physicians (who will not be blinded to treatment condition ["care provider"]) .
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Experimental): Dose of 25 mg daily that may be titrated up to 50 mg daily, if tolerated and will receive treatment as usual for obstructive sleep apnea.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo and will receive treatment as usual for obstructive sleep apnea.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — If tolerated and serum potassium <5.0 meq/L, the dose will be increased to 50 mg (2 pills) after 4 weeks. If serum potassium is >5.0 but less than 5.5 or creatinine >4.0 mg/dL, the dose will be adjusted to 25 mg every other day; if potassium levels ≥5.5 in a non-hemolyzed blood sample, the medication will be discontinued.
  Arms: Spironolactone
Drug: Placebo — Subjects assigned to the placebo group will take one pill for the first 4 weeks and a second pill for the remaining 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether Spironolactone can improve the severity of obstructive sleep apnea and improve cardiovascular biomarkers in people who are not regularly using their Positive Airway Pressure (PAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than or equal to 30
* Diagnosis of moderate to severe OSA via diagnostic polysomnography (AHI≥15) or home sleep apnea test (respiratory event index (REI)≥15).
* Diagnosis of cardiovascular disease
* Meet criteria for hypertension (minimum systolic blood pressure ≥ 140 but <180)
* Prescribed PAP therapy but non-adherent (failure to use PAP for at least 4 hours per night on minimum 5/7 nights per week on average over a one-month period)

Exclusion Criteria:

* Diagnosis of congestive heart failure; resistant hypertension; hepatic disease; Addison's disease; cancer; or recent (past 3 months) myocardial infarction, or stroke
* Diagnosis of central sleep apnea
* Patients who are not using PAP at all (untreated) or using another form of treatment for OSA
* Currently taking, recent trial (past month), or allergy for spironolactone
* Severe respiratory disease (e.g., diagnosis of chronic obstructive pulmonary disease, uncontrolled asthma)
* History of leukopenia and/or thrombocytopenia
* Current use of another potassium sparing diuretic (e.g., amiloride or eplerenone)
* Current use of lithium, barbiturates, narcotics, muscle relaxants, pressor amines, or cholestyramine
* Patients who plan to have surgery during the time period of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in apnea-hypopnea index (AHI) | Day 0, Day 84
  AHI is obtained from polysomnography studies

SECONDARY OUTCOMES:
Change in minimum oxygen saturation (SaO2) | Day 0, Day 84
  Oxygen saturation is obtained from polysomnography studies
Change in Inflammatory biomarker | Day 0, Day 84
  Biomarkers of interest will be obtained via blood draws. Markers of interest: Interleukin 6 protein (IL-6), Tumor necrosis factor alpha (TNF α), High Sensitivity C-Reactive Protein, Brain Natriuretic Peptide (BNP), and procollagen 1 and 3.
Change in Diurnal blood pressure | Day 0, Day 84
  Measured using SPRINT methods; Seated blood pressure is measured after a rest period using an automated device or manual devices if necessary. The preferred method is the automated device. Both systolic and diastolic blood pressure will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Louise O'Brien, PhD, Principal Investigator — University of Michigan; Bertram Pitt, MD, Principal Investigator — University of Michigan; J. Todd Arnedt, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The study team does not have plans to actively share data, however, they are open to collaboration following contact with the investigator.